CLINICAL TRIAL: NCT01629719
Title: STUDY PHASE III COMPARISON OF SUPERIORITY, OPEN WITH BLIND APPRAISER, TO EVALUATE THE EFFICACY AND SAFETY OF BARIUM SULPHATE 66.7% W / V (OPTI-BAR) COMPARED TO PROCEEDINGS IN INERT RADIOLOGICAL EXAMINATIONS FOR THE DIAGNOSIS OF DISEASES FOR IMAGE THE TRATOGASTROINTSTINAL.
Brief Title: Study Phase III Comparison of Superiority, Open With Blind Appraiser, to Evaluate the Efficacy and Safety of Barium Sulphate 66.7% With V (OPTI-BAR) Compared to Proceedings in Inert Radiological Examinations for the Diagnosis of Diseases for Image the Tratogastrointstinal
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Alko Do Brasil Industria e Comercio Ltda (Industry)
Responsible Party: Sponsor
Other Study IDs: ALK 002-001
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: X-ray Examinations of the Gastrointestinal Tract

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Phase III clinical study, two samples, with assessor blind for the purpose of evaluating the efficacy and safety of the superiority of the use of barium sulphate 66.7% w/v (Opti-bar) as a contrast X-ray (X-ray).

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 who need x-rays gastrointestinal tract with contrast;
* Healthy patient, ambulatory;
* Willingness to comply with the requirements of the study after signing an informed consent and (hit).

Exclusion Criteria:

* Pregnant or lactating women;
* Patients allergic to barium sulfate, latex rubber or simethicone;
* Patients who have asthma, eczema, cystic fibrosis, heart disease, high blood pressure, rectal cancer, colostomy, obstruction in the stomach or intestines, pseudotumor cerebri, blocking stomach or intestinal disease, Hirsch or pseudotumor cerebri;
* Patients who have recently undergone a rectal biopsy or surgery or a recent history of drilling into your esophagus, stomach or intestines; Patients who have already participated in another clinical protocol in the last six months;
* Other clinical criteria that in the opinion of the study investigator could compromise the welfare of the patient or interfere with the results expected from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women over 18 years.
Sampling Method: Probability Sample
Enrollment: 73 (Estimated)
Dates: Start 2012-06